CLINICAL TRIAL: NCT01401075
Title: Prospective Controlled Randomized Comparative Study About Quality of Life (QoL), Immunomodulation and Safety of Adjuvant Mistletoe Treatment in Patients With Gastric Carcinoma Receiving Chemotherapy After Operation
Brief Title: RCT With Adjuvant Mistletoe Treatment in Gastric Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abnoba Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AB-AVQ20-1.0
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2011-07

CONDITIONS: Gastric Cancer
Keywords: Quality of Life; QoL; EORTC QLQ-C30; EORTC QLQ-STO22; 5-FU; Viscum album
MeSH Terms: conditions — Stomach Neoplasms | interventions — doxifluridine; 3,4-dihydroxybenzohydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- doxifluridine (Active Comparator): oral chemotherapy with the 5-FU prodrug doxifluridine
  Interventions: Drug: doxifluridine
- doxifluridine + mistletoe extract (Experimental): oral chemotherapy with the 5-FU prodrug doxifluridine + mistletoe extract as subcutaneous injection
  Interventions: Drug: mistletoe extract; Drug: doxifluridine

INTERVENTIONS:
Drug: mistletoe extract — subcutaneous injections thrice weekly with 1 ml in 4 increasing doses
  Other Names: abnobaVISCUM Quercus 0.02 mg; abnobaVISCUM Quercus 0.2 mg; abnobaVISCUM Quercus 2 mg; abnobaVISCUM Quercus 20 mg
  Arms: doxifluridine + mistletoe extract
Drug: doxifluridine — 600 - 900 mg per day orally, depending on weight and status of the patient
  Other Names: Didox

SUMMARY:
Evaluation of safety and efficacy of a standardized mistletoe extract (abnobaVISCUM® Quercus, aVQ) in patients with gastric cancer receiving oral chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* postoperative UICC stage Ib/II gastric carcinoma
* indication for oral chemotherapy with doxifluridine
* ECOG performance status 0 or 1
* normal liver and kidney function

Exclusion Criteria:

* inability to answer the QoL scales
* concomitant therapy with steroids or biological response modifiers
* individual hypersensitivity to mistletoe preparations
* pregnancy or lactating
* participation in another clinical trial

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 24 weeks
  EORTC Quality of Life Questionnaires:
  1. QLQ-C30
  2. QLQ-STO22

SECONDARY OUTCOMES:
Immunomodulation | 24 weeks
  1. cytokine levels (TNF-alpha and interleukin-2)
  2. lymphocyte subsets (CD 16+/CD56+ and CD 19+)
Safety and tolerability | 24 weeks
  1. differential blood count
  2. liver functions tests
  3. adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Sik Kim, Professor, Principal Investigator — ASAN Medical Center, Seoul
Locations (1):
- ASAN Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Kim KC, Yook JH, Eisenbraun J, Kim BS, Huber R. Quality of life, immunomodulation and safety of adjuvant mistletoe treatment in patients with gastric carcinoma - a randomized, controlled pilot study. BMC Complement Altern Med. 2012 Oct 3;12:172. doi: 10.1186/1472-6882-12-172. PMID 23033982